CLINICAL TRIAL: NCT06294431
Title: Radicle Clarity™ 24: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Cognitive Function and Related Health Outcomes
Brief Title: Radicle Clarity 24: A Study of Health and Wellness Products on Cognitive Function and Related Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-P-2406
Record Dates: First submitted 2024-02-21; First posted 2024-03-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Function

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their gender assigned at birth and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (17):
- Placebo Control 1 (Placebo Comparator): Clarity Product Form 1 - control
  Interventions: Dietary Supplement: Placebo Control Form 1
- Active Product 1.1 (Experimental): Clarity Product Form 1 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 1.1 Usage
- Placebo Control 2 (Placebo Comparator): Clarity Product Form 2 - control
  Interventions: Dietary Supplement: Placebo Control Form 2
- Active Product 2.1 (Experimental): Clarity Product Form 2 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 2.1 Usage
- Placebo Control 3 (Placebo Comparator): Clarity Product Form 3 - control
  Interventions: Dietary Supplement: Placebo Control Form 3
- Active Product 3.1 (Experimental): Clarity Product Form 3 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 3.1 Usage
- Active Product 3.2 (Experimental): Clarity Product Form 3 - active product 2
  Interventions: Dietary Supplement: Clarity Active Study Product 3.2 Usage
- Placebo Control 4 (Placebo Comparator): Clarity Product Form 4 - control
  Interventions: Dietary Supplement: Placebo Control Form 4
- Active Product 4.1 (Experimental): Clarity Product Form 4 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 4.1 Usage
- Placebo Control 5 (Placebo Comparator): Clarity Product Form 5 - control
  Interventions: Dietary Supplement: Placebo Control Form 5
- Active Product 5.1 (Experimental): Clarity Product Form 5 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 5.1 Usage
- Active Product 5.2 (Experimental): Clarity Product Form 5 - active product 2
  Interventions: Dietary Supplement: Clarity Active Study Product 5.2 Usage
- Placebo Control 6 (Placebo Comparator): Clarity Product Form 6 - control
  Interventions: Dietary Supplement: Placebo Control Form 6
- Active Product 6.1 (Experimental): Clarity Product Form 6 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 6.1 Usage
- Placebo Control 6.1.0 (Placebo Comparator): Clarity Product 6.1.0 - control
  Interventions: Dietary Supplement: Placebo Control 6.1.0
- Active Product 6.1.1 (Experimental): Clarity Product 6.1.1 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 6.1.1 Usage
- Active product 6.1.2 (Experimental): Clarity Product 6.1.2
  Interventions: Dietary Supplement: Clarity Active Study Product 6.1.2 Usage

INTERVENTIONS:
Dietary Supplement: Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Clarity Active Study Product 1.1 Usage — Participants will use their Radicle Clarity Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Placebo Control Form 2 — Participants will use their Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Clarity Active Study Product 2.1 Usage — Participants will use their Radicle Clarity Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Placebo Control Form 3 — Participants will use their Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Clarity Active Study Product 3.1 Usage — Participants will use their Radicle Clarity Active Study Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1
Dietary Supplement: Clarity Active Study Product 3.2 Usage — Participants will use their Radicle Clarity Active Study Product 3.2 as directed for a period of 6 weeks.
  Arms: Active Product 3.2
Dietary Supplement: Placebo Control Form 4 — Participants will use their Placebo Control Form 4 as directed for a period of 6 weeks.
  Arms: Placebo Control 4
Dietary Supplement: Clarity Active Study Product 4.1 Usage — Participants will use their Radicle Clarity Active Study Product 4.1 as directed for a period of 6 weeks.
  Arms: Active Product 4.1
Dietary Supplement: Placebo Control Form 5 — Participants will use their Placebo Control Form 5 as directed for a period of 6 weeks.
  Arms: Placebo Control 5
Dietary Supplement: Clarity Active Study Product 5.1 Usage — Participants will use their Radicle Clarity Active Study Product 5.1 as directed for a period of 6 weeks.
  Arms: Active Product 5.1
Dietary Supplement: Clarity Active Study Product 5.2 Usage — Participants will use their Radicle Clarity Active Study Product 5.2 as directed for a period of 6 weeks.
  Arms: Active Product 5.2
Dietary Supplement: Placebo Control Form 6 — Participants will use their Placebo Control Form 6 as directed for a period of 6 weeks.
  Arms: Placebo Control 6
Dietary Supplement: Clarity Active Study Product 6.1 Usage — Participants will use their Radicle Clarity Active Study Product 6.1 as directed for a period of 6 weeks.
  Arms: Active Product 6.1
Dietary Supplement: Placebo Control 6.1.0 — Participants will use their Placebo Control 6.1.0 as directed for a period of 6 weeks.
  Arms: Placebo Control 6.1.0
Dietary Supplement: Clarity Active Study Product 6.1.1 Usage — Participants will use their Radicle Clarity Active Study Product 6.1.1 as directed for a period of 6 weeks.
  Arms: Active Product 6.1.1
Dietary Supplement: Clarity Active Study Product 6.1.2 Usage — Participants will use their Radicle Clarity Active Study Product 6.1.2 as directed for a period of 6 weeks.
  Arms: Active product 6.1.2

SUMMARY:
A randomized, double-blind, placebo-controlled direct-to-consumer study of health and wellness products on cognitive function and related health outcomes

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) endorse a desire for better concentration, (2) have the opportunity for meaningful improvement (at least 20%) in their primary health outcome, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic, there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities. Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Endorses better concentration or cognitive function (fewer feelings of brain fog) as a primary desire
* Has the opportunity for at least 20% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety lak
* Reports a diagnosis or cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients. NYHA (New York Heart Association) Class Ill or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients. Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOls (monoamine oxidase inhibitors), or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s)
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4794 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | 6 weeks
  Mean difference in cognition function score as assessed by Patient Reported Outcome Measurement System (PROMIS) Cognitive Function Short Form 8A (scale 8-40; where the higher scores correspond to greater cognitive function)

SECONDARY OUTCOMES:
Change in fatigue | 6 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Change in sleep-related impairment | 6 weeks
  Mean difference in sleep-related impairment score as assessed by PROMIS Sleep-Related Impairment 4A (scale 4-20; with higher scores corresponding to greater sleep-related impairment)
Minimal clinical importance difference (MCID) in cognitive function | 6 weeks
  Likelihood of achieving a MCID in cognitive function, as measured by PROMIS Cognitive Function Short Form 8A (scale 8-40; where the higher scores correspond to greater cognitive function)

OTHER OUTCOMES:
Change in mood (emotional distress-depression) | 6 weeks
  Mean difference in mood score as assessed by PROMIS Depression 4A (scale 4-20; where higher scores correspond to more severe depression)
Change in concentration of at-home (direct-to-consumer) specimen assays either saliva, blood or stool | 6 weeks
  Mean difference in specimen assays as surrogates and/or markers for health outcomes. (Optional; among consented participants only) Potentially include saliva (IgG, cytokines, DHEA-S, Estradiol, Progesterone, Testosterone, Cortisol, Melatonin, CRP) blood (1 drop) (Cortisol, Homocysteine, Ferritin, TSH, HbA1c, Insulin, Vitamin D, DHEA-S, Testosterone, Estradiol, FSH, Total Cholesterol, HDL, LDL, Triglycerides, ApoA1, ApoB). Stool (microbial diversity).

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com